CLINICAL TRIAL: NCT07258979
Title: A Multicenter, Open-label, Phase Ib/II Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of YL201 Combined With Toripalimab, With or Without Cisplatin, in Subjects With Recurrent or Metastatic Nasopharyngeal Carcinoma.
Brief Title: A Study of YL201 in Combination With Toripalimab and With or Without Cisplatin in Nasopharyngeal Carcinoma.
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MediLink Therapeutics (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YL201-CN-105-02
Record Dates: First submitted 2025-11-17; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Recurrent or Metastatic Nasopharyngeal Carcinoma
Keywords: YL201; recurrent or metastatic nasopharyngeal carcinoma; Toripalimab
MeSH Terms: conditions — Recurrence; Nasopharyngeal Carcinoma | interventions — toripalimab; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose Exploration (Part 1) (Experimental): To evaluate the safety and efficacy of YL201 combined with Toripalimab in subjects with recurrent or metastatic nasopharyngeal carcinoma
  Interventions: Drug: YL201; Drug: Toripalimab
- Dose Exploration (Part 2) (Experimental): To evaluate the safety and efficacy of YL201 combined with Toripalimab with/without Cisplatin in subjects with recurrent or metastatic nasopharyngeal carcinoma.
  Interventions: Drug: YL201; Drug: Toripalimab; Drug: Cisplatin

INTERVENTIONS:
Drug: YL201 — YL201 will be administered as an IV infusion
Drug: Toripalimab — Toripalimab will be administered as an IV infusion
Drug: Cisplatin — Cisplatin will be administered as an IV infusion
  Arms: Dose Exploration (Part 2)

SUMMARY:
This is a multicenter, open-label, Phase Ib/II study conducted in China to evaluate the safety, efficacy, and pharmacokinetic (PK) characteristics of YL201 combined with Toripalimab (doublet regimen) or YL201 combined with Toripalimab and Cisplatin (triplet regimen) in subjects with recurrent or metastatic nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign a written informed consent form (ICF).
2. Aged ≥18 years and ≤75 years, male or female.
3. ECOG performance status score of 0 or 1.
4. Life expectancy ≥ 3 months.
5. Disease and treatment history:

   1. Histologically or cytologically confirmed recurrent or metastatic nasopharyngeal carcinoma that is not amenable to curative treatment.
   2. Patients with newly diagnosed advanced nasopharyngeal carcinoma, categorized as Stage IV according to the 9th Edition of the American Joint Committee on Cancer (AJCC) Staging System; or those with recurrent nasopharyngeal carcinoma deemed unsuitable for local treatment
   3. Metastatic or recurrent patients who are systemic treatment naïve.
6. At least one measurable lesion according to RECIST v1.1.
7. Adequate organ function.

Exclusion Criteria:

1. History of other malignant tumors within 5 years prior to the first dose of study drug. Subjects who have been cured of other tumors by local therapy, such as basal cell carcinoma, squamous cell carcinoma of skin, bladder cancer in situ, cervical carcinoma in situ, or breast cancer in situ, are not excluded.
2. Patients with brainstem metastases, leptomeningeal metastases, spinal cord metastases, or spinal cord compression.
3. Patients with severe, uncontrolled cardiovascular disease.
4. Patients with concomitant pulmonary disease resulting in clinically severe impairment of respiratory function.
5. History of interstitial lung disease (ILD) or non-infectious pneumonitis requiring corticosteroid therapy, OR current ILD or non-infectious pneumonitis.
6. Prior treatment with a B7-H3 targeted therapy (including antibodies, antibody-drug conjugates [ADCs], CAR-T cells, and other agents), or with a topoisomerase I inhibitor or an ADC containing a topoisomerase I inhibitor payload.
7. Prior treatment with a PD-(L)1 inhibitor (including antibodies, antibody-drug conjugates [ADCs], CAR-T cells, and other agents).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing Dose-limiting toxicities (DLTs) | Approximately within 36 months
Number of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) | Approximately within 36 months
Progression-Free Survival (PFS) as assessed by RECIST v1.1 | Approximately within 36 months

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Approximately within 36 months
Disease Control Rate (DCR) | Approximately within 36 months
Time to Response (TTR) | Approximately within 36 months
Duration of Response (DoR) | Approximately within 36 months
Overall survival(OS) | Approximately within 36 months
Incidence of anti-drug antibodies (ADA) to YL201 (and to Toripalimab, if necessary) | Approximately within 36 months
Characterize the PK parameter AUC of YL201 and its metabolites, if applicable | Approximately within 36 months
Characterize the PK parameter Cmax of YL201 and its metabolites, if applicable | Approximately within 36 months
Characterize the PK parameter Ctrough of YL201 and its metabolites, if applicable | Approximately within 36 months
Characterize the PK parameter t1/2 of YL201 and its metabolites, if applicable | Approximately within 36 months

CONTACTS AND LOCATIONS:
Locations (20):
- China (20):
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Zhangzhou Municiple Hospital of Fujian Province, Zhangzhou, Fujian
  - Dongguan People's Hospital, Dongguan, Guangdong
  - Affiliated Cancer Hospital and Institute of Guangzhou Medical University, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangdong Pharmaceutical University, Guangzhou, Guangdong
  - Jiangmen Central Hospital, Jiangmen, Guangdong
  - Yuebei People's Hospital, Shaoguan, Guangdong
  - The Second Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - The First Affiliated Hospital of Hainan Medical University, Haikou, Hainan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No